CLINICAL TRIAL: NCT01198769
Title: Immunogenicity, Reactogenicity and Safety Study of GlaxoSmithKline (GSK) Biologicals' Oral Live Attenuated Human Rotavirus (HRV) Vaccine in Healthy Taiwanese Infants Who Received Hepatitis B Immunoglobulin After Birth.
Brief Title: Immunogenicity and Safety Study of Rotarix TM in Taiwanese Infants Who Received Hepatitis B Immunoglobulin After Birth.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 114351
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Results first posted 2012-04-17 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2016-09

CONDITIONS: Infections, Rotavirus
Keywords: Human rotavirus vaccine
MeSH Terms: conditions — Rotavirus Infections

ARMS (1):
- Rotarix Group (Experimental): subjects received 2 oral doses of Rotarix™ vaccine at 2 and 4 months of age.
  Interventions: Biological: Rotarix TM

INTERVENTIONS:
Biological: Rotarix TM — Oral, 2 doses

SUMMARY:
The purpose of this study is to assess immunogenicity and safety of Rotarix TM when administered in healthy Taiwanese infants (aged 6 to 12 weeks at the time of first vaccination) who received Hepatitis B immunoglobulin after birth.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that parent(s)/Legally Acceptable Representative(s) can and will comply with the requirements of the protocol.
* A male or female between, and including, 6 and 12 weeks of age at the time of the first vaccination.
* Written informed consent obtained from the parent(s)/Legally Acceptable Representative(s) of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Infants who have received a previous dose of hepatitis B immunoglobulin after birth.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs with the exception of Hepatitis B immunoglobulin since birth. Child is unlikely to remain in the study area for the duration of the study.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days of the first dose of vaccine.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Previous vaccination against rotavirus.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness.
* Acute disease and/or fever at the time of enrolment.
* Administration of immunoglobulins (with the exception of HBIG) and/or any blood products since birth or planned administration during the study period.
* Gastroenteritis within 7 days preceding the study vaccine administration.
* Previous confirmed occurrence of Rotavirus gastroenteritis.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2010-11-11; Primary Completion 2011-04-18 (Actual); Study Completion 2011-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Lu CY, Chang LY, Shao PL, Suryakiran PV, Han HH, Huang LM. Immunogenicity, reactogenicity, and safety of a human rotavirus vaccine, Rotarix, in Taiwanese infants who received a dose of hepatitis B immunoglobulin after birth. J Formos Med Assoc. 2013 Sep;112(9):574-7. doi: 10.1016/j.jfma.2012.11.016. Epub 2013 Jan 3. PMID 24079716
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 114351 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114351 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114351 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114351 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114351 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114351 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114351 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rotarix Group
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rotarix Group
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 8.9 (0.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted Subjects for Serum Anti-rotavirus Immunoglobulin A (IgA) Antibody.
Description: Seroconversion is defined as the appearance of IgA antibody concentration equal to or above (≥) 20 Units per millilitre (U/mL) in the serum of subjects who were seronegative before vaccination. A seronegative subject is a subject with anti-rotavirus IgA antibody concentration below (<) 20 U/mL.
Time Frame: 2 months post-Dose 2 (at study Month 4)
Population: The According-To-Protocol cohort for immunogenicity included subjects who received Hepatitis B immunoglobulin after birth, who were seronegative for serum anti-RV IgA antibody at Day 0, who complied with vaccination schedule for the Rotarix vaccine, who had no RV other than the vaccine strain in gastroenteritis stool sample up to Month 4.
Measure: Number; unit: Subjects
Arm/Group | Rotarix Group
Number analyzed (Participants) | 15
Subjects | 15

2. Secondary Outcome: Serum Anti-rotavirus IgA Antibody Concentrations.
Description: Concentrations were expressed as geometric mean antibody concentration in units per millilitre (U/mL), calculated on all subjects.
Time Frame: 2 months post-Dose 2 (at study Month 4)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | Rotarix Group
Number analyzed (Participants) | 15
U/mL | 254.7 [145.0 to 447.7]

3. Secondary Outcome: Number of Subjects Reporting Solicited General Symptoms.
Description: Solicited general symptoms assessed were cough, diarrhoea, irritability, loss of appetite, temperature (any temperature was defined as a tympanic on rectal setting temperature ≥ 38.0 degrees Celsius) and vomiting.
Time Frame: During the 8-day (Days 0-7) post-vaccination period
Population: The Total vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | Rotarix Group
Number analyzed (Participants) | 15
Subjects
  Cough | 6
  Diarrhoea | 1
  Irritability | 11
  Loss of appetite | 10
  Temperature (Tympanic on rectal seting (>=38.0°C)) | 5
  Vomiting | 2

4. Secondary Outcome: Number of Subjects With Rotavirus (RV) Present in the Gastroenteritis (GE) Stool Sample.
Description: RV was not identified in the one GE stool sample collected in the study. Two subjects reported GE episode between vaccination Dose 1 and before vaccination Dose 2. For one of them, GE stool sample was not collected and for the other subject no RV was identified in the GE stool sample.
  GE symptoms were defined as diarrhoea with or without vomiting. A GE stool sample was collected as soon as possible after the illness began by the parent/guardian of the subject. Presence of RV antigen was detected by Enzyme-linked immunosorbent assay (ELISA).
Time Frame: From Day 0 (first vaccine dose) to study Month 4 (2 months post-Dose 2)
Population: The Total vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | Rotarix Group
Number analyzed (Participants) | 15
Subjects | 0

5. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs).
Description: An unsolicited adverse event is any adverse event (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Within the 31-day (Days 0-30) follow-up period after vaccination
Population: The Total vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | Rotarix Group
Number analyzed (Participants) | 15
Subjects | 4

6. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs).
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects.
Time Frame: During the entire study period (from Dose 1 at Day 0 up to Month 4)
Population: The Total vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | Rotarix Group
Number analyzed (Participants) | 15
Subjects | 1

ADVERSE EVENTS:
Time Frame: SAEs: During the entire study period (from Dose 1 at Day 0 up to Month 4). Unsolicited AEs: Within the 31-day (Days 0-30) follow-up period after vaccination. Solicited general symptoms: During the 8-day (Days 0-7) post-vaccination period
Arm/Group | Rotarix Group
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rotarix Group (N=15)
Bronchiolitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rotarix Group (N=15)
Eczema (Skin and subcutaneous tissue disorders) | 2
Bronchiolitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Cough (General disorders) | 6
Diarrhoea (General disorders) | 1
Irritability (General disorders) | 11
Loss of appetite (General disorders) | 10
Temperature (General disorders) | 5
Vomiting (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.